CLINICAL TRIAL: NCT04392557
Title: Comparison of Anti-inflammatory Status Linked to Atherosclerosis Formation/Progression Among Diabetes Mellitus Type 2 Patients Under Combined Pharmacological Therapy
Brief Title: Anti-inflammatory Status in DM2 Treated Patients
Acronym: INF-DM2-Ther
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, Principal investigator, University of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Inflammation-DM2
Record Dates: First submitted 2020-05-04; First posted 2020-05-19 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Pioglitazone

STUDY DESIGN:
Intervention Model Description: single center single blind study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- metformin/alogliptin (Active Comparator): metformin/alogliptin (850 mg/12.5 mg or 1000 mg/12.5 mg every 12 hours) for 12 months
  Interventions: Drug: Metformin / alogliptin Oral Product
- metformin/pioglitazone (Active Comparator): metformin/pioglitazone (850 mg/15 mg every 12 hours) for 12 months
  Interventions: Drug: Metformin / Pioglitazone Pill
- triple therapy (Active Comparator): metformin/pioglitazone (850 mg/15 mg every 12 hours)+alogliptin (12.5 mg every 12 hours) for 12 months
  Interventions: Drug: Metformin / alogliptin Oral Product; Drug: Metformin / Pioglitazone Pill; Drug: triple therapy

INTERVENTIONS:
Drug: Metformin / alogliptin Oral Product — 850 or 1000 mg/ 12.5 mg every 12 hours for 12 months
  Arms: metformin/alogliptin; triple therapy
Drug: Metformin / Pioglitazone Pill — (850 mg/15 mg every 12 hours) for 12 months
  Arms: metformin/pioglitazone; triple therapy
Drug: triple therapy — Metformin / Alogliptin/ Pioglitazone
  Arms: triple therapy

SUMMARY:
Diabetes mellitus Type 2 (DMT2) - a progressive insulin secretory defect on the background of insulin resistance - is one of the major risk factors for atherosclerosis, an inflammatory disease of the arterial wall, in which leukocytes and oxidized lipoproteins accumulate leading to formation of fatty streaks and atherosclerotic plaques. Atherosclerosis accounts for more than 600,000 deaths annually in the U.S. mainly due to acute myocardial infarction and stroke. Pharmacological therapy of DMT2 includes several drugs used as monotherapy, although combination therapy between metfomin plus thiazolidinediones (TZD) and/or dipeptidyl-peptidase 4 inhibitors (DPP4I) plus TDZ, may delay atherosclerosis progression even if the molecular mechanisms are not clear. Even if normoglycemia is achieved, DMT2 patients still displayed a higher risk for developing atherosclerosis suggesting that other mechanisms of the inflammatory status are involved

DETAILED DESCRIPTION:
Diabetes mellitus Type 2 (DMT2) - a progressive insulin secretory defect on the background of insulin resistance - is one of the major risk factors for atherosclerosis, an inflammatory disease of the arterial wall, in which leukocytes and oxidized lipoproteins accumulate leading to formation of fatty streaks and atherosclerotic plaques. Atherosclerosis accounts for more than 600,000 deaths annually in the U.S. mainly due to acute myocardial infarction and stroke. Pharmacological therapy of DMT2 includes several drugs used as monotherapy, although combination therapy between metfomin plus thiazolidinediones (TZD) and/or dipeptidyl-peptidase 4 inhibitors (DPP4I) plus TDZ, may delay atherosclerosis progression even if the molecular mechanisms are not clear . Even if normoglycemia is achieved, DMT2 patients still displayed a higher risk for developing atherosclerosis suggesting that other mechanisms of the inflammatory status are involved

ELIGIBILITY:
Inclusion Criteria:

* DMT2 patients were enrolled in presence of

  1. Age >35 and <75 years old
  2. Uncontrolled diabetes during treatment (glycosylated hemoglobin (HbA1c) > 75 mmol/mol )
  3. Combined therapy at least by 6 months.

Exclusion Criteria:

1. HbA1c < 75 mmol/mol (9%);
2. History of drug abuse or alcohol abuse, averaging more than 30 gm/day (3 drinks per day) in the previous 10 years, or history of alcohol intake averaging greater than 10 gm/day (1 drink per day: 7 drinks per week) in the previous one year;
3. Estimated glomerular filtration rate (GFR) <30 ml/min (according to MDRD formula)
4. .Liver Failure
5. Recent history of Heart stroke, systemic infections, dehydration, lactic acidosis
6. Heart failure (NYHA I - IV)
7. Active bladder cancer or history of bladder cancer
8. macroscopic haematuria of unidentified nature
9. hypersensitivity to drug used (metformin, alogliptin, pioglitazone)
10. breastfeeding

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-06-20 (Estimated)

PRIMARY OUTCOMES:
inflammatory miRNA | 12 months
  Change from Baseline at 12 months
side effects | 12 months
  statistically significant difference (P<0.05) in the development of side effects between the groups, recorded using the Naranjo adverse drug reactions scale

SECONDARY OUTCOMES:
body weight | 12 months
  effects of each treatment on body mass index (kg/m^2) (as indirect indexes of systemic inflammation and visceral adiposity).
Waist values | 12 months
  effects of each treatment on waist values (cm) (as indirect indexes of systemic inflammation and visceral adiposity).
drug interaction | 12 months
  statistically significant difference (P<0.05) in the development of drug-drug interactions, recorded using the DIPS scale
Fasting blood glucose | 12 months
  effects of each treatment on fasting blood glucose (mg/dL) (as indexes of glucose metabolism);
HbA1c levels | 12 months
  effects of each treatment on HbA1c levels (percent) (as indexes of glucose metabolism);
liver function | 12 months
  alanine aminotransferase, aspartate aminotransferase, gamma glutamyl-transpeptidase levels, and total bilirubin levels (expressed as mg/dL) (as indexes of liver function).
cell count | 12 months
  effects of each treatment on white blood cell count expressed as cell/mm3 (as direct index of systemic inflammation)
lipid metabolism/atheroscelorisis | 12 months
  total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides levels (expressed as mg/dL) (as direct indexes of lipid metabolism and atheroscelorisis).

CONTACTS AND LOCATIONS:
Locations (1):
- ASP Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No